CLINICAL TRIAL: NCT03967977
Title: A Phase 3, Multi-center, Randomized, Double-Blind, Placebo-Controlled Study of Either Cisplatin or Carboplatin +Gemcitabine + Tislelizumab Compared With Either Cisplatin or Carboplatin + Gemcitabine + Placebo as First-line Treatment for Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Study of Tislelizumab in Combination With Chemotherapy Compared to Chemotherapy Alone for Participants With Urothelial Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-A317-310; CTR20190543 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — tislelizumab; Cisplatin; Gemcitabine; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab in combination with chemotherapy (Active Comparator): Tislelizumab: Day 1 of each 21-day cycle, to be administered until Progressive Disease or intolerable toxicity Cisplatin: Day 1 or Day 2 of each 21-day cycle, to be administered up to 6 cycles Carboplatin: Day 1 or Day 2 of each 21-day cycle, to be administered up to 6 cycles Gemcitabine: Days 1 and 8 of each 21-day cycle, to be administered up to 6 cycles
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Carboplatin
- Placebo in combination with chemotherapy (Placebo Comparator): Placebo: Day 1 of each 21-day cycle, to be administered until Progressive Disease or intolerable toxicity Cisplatin: Day 1 or Day 2 of each 21-day cycle, to be administered up to 6 cycles Carboplatin: Day 1 or Day 2 of each 21-day cycle, to be administered up to 6 cycles Gemcitabine: Days 1 and 8 of each 21-day cycle, to be administered up to 6 cycles
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — 200 mg administered Intravenously (IV) as specified in the treatment arm
  Other Names: BGB-A317
  Arms: Tislelizumab in combination with chemotherapy
Drug: Placebo — Tislelizumab placebo to match
  Arms: Placebo in combination with chemotherapy
Drug: Cisplatin — 70 mg/m2 administered IV as specified in the treatment arm
Drug: Gemcitabine Hydrochloride — 1000 mg/m2 administered IV as specified in the treatment arm
Drug: Carboplatin — Area Under the Curve (AUC) 4.5 administered IV as specified in the treatment arm

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase 3 study designed to compare the efficacy and safety of tislelizumab + either cisplatin or carboplatin + gemcitabine versus placebo+ either cisplatin or carboplatin + gemcitabine in approximately 420 participants with locally advanced or metastatic urothelial carcinoma who have not received prior systemic therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged 18 to 75 years on the day of signing the Informed Consent Form (ICF)
2. Histologically confirmed, inoperable, locally advanced, or metastatic urothelial cancer (UC)
3. Must be eligible to receive cisplatin or carboplatin in the investigator's judgment
4. Have had no prior systemic chemotherapy for locally advanced or metastatic UC
5. Must be able to provide fresh or archival tumor tissues with an associated pathological report.
6. Must have evaluable disease (either measurable or non-measurable) as defined per RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
8. Adequate organ function before randomization:

Key Exclusion Criteria:

1. Received prior therapies targeting PD-1, PD-L1, PD-L2, CTLA4, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
2. Any approved anticancer therapy within 28 days before randomization.
3. Active leptomeningeal disease or uncontrolled, untreated brain metastasis
4. Participants with uncontrolled hypercalcemia
5. Participants with active autoimmune diseases or history of autoimmune diseases that may relapse
6. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled diseases
7. A known history of HIV infection.
8. Prior allogeneic stem cell transplantation or organ transplantation.
9. History of severe hypersensitivity reactions to other monoclonal antibodies. 10．History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in the Intent to Treat (ITT) set | From first randomization up to 3.5 years, approximately

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 in ITT | From first randomization up to 3.5 years, approximately
  the proportion of participants who had Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST v1.1 in the ITT Analysis Set
Duration of response (DOR) | From first randomization up to 3.5 years, approximately
  the time from the first occurrence of a documented objective response to documented Progressive Disease (PD), or death from any cause, whichever occurs first, as determined by the investigator per RECIST v1.1 in the ITT Analysis Set
Progression-free survival (PFS) | From first randomization up to 3.5 years, approximately
  the time from randomization to the first objectively documented PD, or death from any cause, whichever occurs first, as determined by the investigator per RECIST v1.1 in the ITT Analysis Set
Overall survival rate at 1 and 2 years for each treatment arm | From first randomization up to 3.5 years, approximately
  the proportion of OS participants at 1 year and 2 years from randomization in the ITT Analysis Set
Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life-Core 30(EORTC QLQC30) | From first randomization up to 3.5 years, approximately
  1) to assess overall health status/Quality of Life with 2 questions which are with range from minimum score 1 as worse outcome and maximum score 7 as higher values represent a better 2) to assess quality of life with 28 questions about Physical functioning, emotional functioning, social functioning etc. which are with range from minimum scores 1 representing as better to maximum scores 4 as worse outcome.
Incidence and severity of treatment-emergent adverse events (AEs) | From first randomization up to 3.5years, approximately
  Incidence and severity of treatment-emergent adverse events (AEs) graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)v5.0
Change from baseline in European Quality of Life 5-Dimension, 5-Level version (EQ-5D-5L) | From first randomization up to 3.5 years, approximately
  to assess health status with 1) 5 questions about Mobility, Self-Care, Usual activities, Pain/Discomfort, Anxiety/Depression which are with 5 options. 2) one question about health status at the day of completing the questionnaire with range from minimum score 0 as worse outcome to maximum scores 100 as higher values represent as better.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD, Principal Investigator — Fudan University
Locations (46):
- China (41):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fifth Medical Center of Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Provincial Wenzhou Hospital of Zhejiang, Wenzhou, Zhejiang
- Taiwan (5):
  - Keelung Chang Gung Memorial Hospital and Loves Lake Branch, Anle Dist
  - Taipei Veterans General Hospital, Beitou Dist
  - Linkou Chang Gung Memorial Hospital, Guishan Dist
  - National Cheng Kung University Hospital, North Dist
  - National Taiwan University Hospital, Zhongzheng Dist

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/